CLINICAL TRIAL: NCT01914406
Title: High-intensity Interval Training Versus Moderate Continuous Training in Heart Transplant Recipients With Impaired Chronotropic Response: A Randomized Controlled Crossover Trial.
Brief Title: High-intensity Interval Training Versus Moderate Continuous Training in Heart Transplant Recipients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christian Dall, Associate professor, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2010 030
Record Dates: First submitted 2013-07-25; First posted 2013-08-02 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Heart Transplant Recipients
Keywords: Heart transplant recipients; Exercise capacity; endothelial function; Quality of life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high intense interval training (Other): Each AIT session consisted a 10 minute warm-up period followed by 16 minutes of interval training consisting of intervals of 4-3-2 and 1 minutes duration at 85-95% of their peak capacity separated by 2-4 min active rest.
  Interventions: Other: high intense interval training
- continuous moderate training (Active Comparator): Continued exercise 45 min.
  Interventions: Other: continuous moderate training

INTERVENTIONS:
Other: high intense interval training — Each AIT session consisted a 10 minute warm-up period followed by 16 minutes of interval training consisting of intervals of 4-3-2 and 1 minutes duration at 85-95% of their peak capacity separated by 2-4 min active rest.
  Arms: high intense interval training
Other: continuous moderate training — Continued exercise 45 min.
  Arms: continuous moderate training

SUMMARY:
The aim of this study was to examine the effects of high intensity aerobic interval training (AIT) versus moderate continuous training (CON) in heart transplant recipients.

DETAILED DESCRIPTION:
Clinically stable heart transplant recipients > 12 month or more after HTx, age > 18 years, willing and capable of giving written informed consent for study participation and anticipated to be able to participate in the study for 12 months were included from the Heart Centre, Rigshospitalet, Copenhagen University Hospital.

Patients were excluded due to unstable condition or postoperative complications, recent severe rejection episodes (>H1R < 3 month), physical disabilities which prevent participation and re-transplantation or multi-organtransplantation.

ELIGIBILITY:
Inclusion Criteria:

-stable Heart transplant recipients > 12 month or more after HTx, age > 18 years,< 80. willing and capable of giving written informed consent for study participation.

Exclusion Criteria:

unstable condition postoperative complications, recent severe rejection episodes (>H1R < 3 month), re-transplantation or multi-organtransplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
VO2peak | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  baseline test before randomization
  1. follow-up after 12 weeks of exercise
  2. follow-up after 5 month washout.
  3. follow-up after second 12 weeks period of exercise.

SECONDARY OUTCOMES:
Endothelial function (endoPAT) | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  After the release of the cuff the hyperemic response was recorded and the reactive hyperemia index (RHI) was calculated automatic independent of operator. (endoPAT)
Quality of Life (QoL)SF-36 | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  SF-36, information on Quality of Life
HADS-a, HADS-d anxiety and depression | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  Symptoms of anxiety and depression measured by the Hospital Anxiety and Depression Scale (HADS).
Bloodsamples/biomarkers. | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  Samples cooled on ice, centrifuged for 10 minutes and the plasma transferred to microtubes and stored at -80°C. Biomarkers analysed at department of biomedicine at University of Copenhagen.
augmentation index (AI), endoPAT | baseline test (inclusion), follow-up 1(3 month), follow-up 2 (8 month), follow-up 3 (11 month).
  Augmentation index (AI)derived from pulse wave analyses and is a measure of arterial stiffness, (EndoPAT).

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Dall, cand.scient, Principal Investigator — Bispebjerg Hospital, Denmark
Locations (1):
- Cardiac Rehabilitation, Bispebjerg University Hospital, Copenhagen, Denmark